CLINICAL TRIAL: NCT03834103
Title: Feasibility Study of a Post-hospitalization Self-rehabilitation Program for Elderly Suffering of Sarcopenia
Acronym: FREESARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-01-2018
Record Dates: First submitted 2019-01-21; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: Self-rehabilitation arm (Other): Self-rehabilitation arm
  Interventions: Behavioral: Self-rehabilitation program and protein supplement

INTERVENTIONS:
Behavioral: Self-rehabilitation program and protein supplement — Participants follow a home-based self-rehabilitation program consisting of the realisation of a set of physical exercises using an elastic band. The exercises have to be performed 3 times a week, and are associated with a protein supplementation.
  The rehabilitation follow-up by the physician is planned once a week, by phone, and with face-to-face appointments at inclusion, 6 weeks and 3 months follow-up.

SUMMARY:
Loss of autonomy among elderly during and after hospitalisation is a well-known problem. Patient suffering of sarcopenia (decreasing in muscle mass and function) are more likely not to recover their previous autonomy.

Studies have shown that physical exercise, especially resistance exercises, is the most efficient known treatment of sarcopenia. Several institution-based rehabilitation programs had been implemented in this purpose.

On the other hand, some studies have shown that home-based self-rehabilitation can be as efficient as institution-based rehabilitation, for example in stroke, cardiac failure and COPD rehabilitation.

The investigators propose to set up a home-based self-rehabilitation program to fight against sarcopenia and hence increasing autonomy among elderly. This study aimed to establish the feasibility of such a program.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or older
* Non-institutionnalised patients
* Patients suffering of sarcopenia during hospitalisation (assessed by the Short Physical Performance Battery, Bio-Impedance analysis and griptest)
* Patients hospitalised in the service of Internal Medicine of Institut Mutualiste Montsouris
* Patients returning at home after hospitalisation
* Patients who gave their written consent
* Patients who benefits from a social security coverage

Exclusion Criteria:

* Patients suffering from a severe medical condition not allowing them to follow a physical exercise program
* Palliative care patients
* Patients without the musculo-squelettic capacity to follow the program : 4/4 on seated postural stability scale ; no motor deficit on lower limb muscular testing ; quadricipital locking when standing
* Patients with severe cognitive disorders (according to MMSE score adapted to socio-cultural level and age)
* Patients who live more than 150 km away
* Patients following specific physiotherapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Feasability of a post-hospitalization self-rehabilitation program for sarcopenic elderly patients | 3 months
  Measured from program adherence using a patient notebook
Feasability of a post-hospitalization self-rehabilitation program for sarcopenic elderly patients | 3 months
  Measured from patient satisfaction using a satisfaction scale
Feasability of a post-hospitalization self-rehabilitation program for sarcopenic elderly patients | 3 months
  Measured from medical time required by phone call

SECONDARY OUTCOMES:
Muscular status evaluation | 3 months
  Change in muscle mass measured with Bio-Impedance analysis
Muscular status evaluation | 3 months
  Performance in muscle mass measured with Short Physical Performance Battery
Muscular status evaluation | 3 months
  Force in muscle mass measured with Grip test
Autonomy degree evaluation | 3 months
  Change in autonomy measured with Barthel Index
Quality of life evaluation | 3 months
  Change in quality of life measured with Médical Outcomes Study Short Form 36

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Mutualiste Montsouris, Paris, France